CLINICAL TRIAL: NCT01360385
Title: Objective Measurement of Retinal Ischemia in Central Retinal Vein Occlusion, and the Effects of Treatment With a Vascular Endothelial Growth Factor Inhibitor.
Brief Title: Retinal Ischemia in Central Retinal Vein Occlusion, and the Effects of Treatment With Intravitreal Ranibizumab
Acronym: LuRVO
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Sindri Traustason, Cand. Scient., Glostrup University Hospital, Copenhagen
Other Study IDs: LuRVO
Record Dates: First submitted 2010-10-28; First posted 2011-05-25 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Central retinal rein occlusion; Retinal oximetry; Oxymap Retinal Oximeter; Visual acuity; Central retinal thickness
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Central Retinal Vein Occlusion: CRVO-patients with planned treatment with intravitreal injections of ranibizumab, who receive three monthly injections of ranibizumab and a 3 month follow-up period, during which ranibizumab injections are provided as needed.

SUMMARY:
Recent studies have shown a remarkably positive effect of 6 monthly injections of Ranibizumab on eyes with CRVO. The disease may cause severe sight threatening complications, partly due to restrictions in blood flow and oxygenation . Although Ranibizumab has been shown affective to reduce oedema of the retina, it is not known whether the drug ameliorates or aggravates restrictions in oxygenation.

The Oxymap oximeter allows a non-invasive measurement of the oxygen saturation in retinal vessels and thus the state of retinal oxygenation.

The primary objective of the study is to evaluate the effects of injections of Ranibizumab on the retinal oxygen saturation in eyes with newly diagnosed central retinal vein occlusion (CRVO),

The secondary objective is to evaluate the effects of injections of Ranibizumab on visual acuity and retinal oedema in eyes with different degree of ischemia.

DETAILED DESCRIPTION:
Background and objectives

The CRUISE study has shown a remarkable positive effect of 6 monthly injections intravitreal Ranibizumab on visual function in eyes with macular edema secondary to CRVO. Eyes with CRVO are at risk of severe complications to retinal ischemia, particularly proliferative retinopathy and neovascular glaucoma. It is not known whether intravitreal anti-VEGF therapy ameliorates or aggravates retinal ischemia and thus the risk of ischemic complications is unknown. Since complications to retinal ischemia take time to develop, and are relatively infrequent, the CRUISE study was not designed, or powered, to investigate the impact of intravitreal anti-VEGF treatment on these complications.

The Oxymap oximeter allows objective non-invasive measurement of the oxygen saturation in retinal vessels and thus the degree of retinal ischemia. The rationale behind the present study is to use this instrument in order to obtain preliminary information on the effects of intravitreal anti-VEGF treatment on retinal ischemia in CRVO eyes without having to wait for ischemic complications to arise in a large study population.

The primary objective of the study is to evaluate the effects of treatment with intravitreal Ranibizumab on the retinal oxygen saturation in eyes with newly diagnosed central retinal vein occlusion (CRVO),

The secondary objective is to evaluate the effects of intravitreal Ranibizumab on visual acuity and central retinal thickness in eyes with different degree of ischemia.

Study design

The research project is a case-series study of CRVO-patients with three monthly injections of Ranibizumab and a 3 month follow-up period, during which Ranibizumab injections are provided as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Central retinal vein occlusion in one eye.
2. Planned treatment with intravitreal injections of Lucentis (ranibizumab)
3. Functional fellow eye.

Exclusion Criteria:

1. Current or previous medical condition that in the opinion of the investigator may confound assessment of study results or put where the study methods may put the patient at risk.
2. Patients who are unable to receive treatment with vascular endothelial growth factor inhibitors.
3. Prior panretinal photocoagulation in the study eye.
4. Prior intraocular surgery in the study eye, other than cataract operation.
5. Any intravitreal injection 6 months prior to study baseline
6. Participation in another clinical study that, in the opinion of the investigator, may confound the assessment of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed central retinal vein occlusion who have planned treatment with intravitreal renibizumab
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Retinal oxygen saturation | 6 months after first injection of ranibizumab.
  Oxygen saturation is measured with the Oxymap Retinal Oximeter, which allows for objective, non-invase oximetry in retinal vessel.
  The outcome measure will be the change in saturation from baseline to 6 months after first injection.

SECONDARY OUTCOMES:
Visual acuity | 6 months after first injection of ranibizumab.
  Visual acuity measured by the ETDRS standard at 4 meters, 2 meters and 1 meter, where applicable.
  The outcome measure will be the mean change in visual acuity, measured in ETDRS letters, from baseline to 6 months after first injection.
Central retinal thickness | 6 months after first injection of ranibizumab.
  Central retinal thickness as measured with optical coherence tomography.
  The outcome measure will be the mean change in central retinal thickness, from baseline to 6 months after first injection.

CONTACTS AND LOCATIONS:
Overall Officials: Morten D la Cour, MD, DMsc, Principal Investigator
Locations (1):
- Department of Ophthalmology, Glostrup Hospital, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Traustason S, la Cour M, Larsen M. Retinal vascular oximetry during ranibizumab treatment of central retinal vein occlusion. Br J Ophthalmol. 2014 Sep;98(9):1208-11. doi: 10.1136/bjophthalmol-2013-304580. Epub 2014 Apr 12. PMID 24729079